CLINICAL TRIAL: NCT05174611
Title: Vitamin D as an Intervention for Improving Quadricep Muscle Strength in Patients After Anterior Cruciate Ligament Reconstruction: A Randomized Double-Blinded, Placebo-Controlled Clinical Trial
Brief Title: Vitamin D to Improve Quadricep Muscle Strength
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020.623
Record Dates: First submitted 2021-11-28; First posted 2022-01-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Quadriceps Muscle Atrophy; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
Keywords: ACL Reconstruction; Vitamin D; Quadricep muscle strength; Quadricep muscle atrophy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into either treatment or placebo groups
Who Masked: Participant, Care Provider
Masking Description: It is double blinded, subject will receive either the supplement or the placebo with same appearance and package. The lot number of the bottle will be used for randomization. And the investigators will ask the manufactory about it at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Subject in treatment group will receive one capsule of 2000IU Vitamin D3 supplement per day with the duration of 16 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo group (Placebo Comparator): Subject in placebo group will receive one capsule of placebo per day which looks exactly same as the Vitamin D3 capsule with the duration of 16 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Subjects will receive 112 capsules with 4 bottles, 28 capsules in each bottle.
  Arms: Treatment group
Other: Placebo — Subjects will receive 112 capsules with 4 bottles, 28 capsules in each bottle.
  Arms: Placebo group

SUMMARY:
Quadriceps muscle strength is one of the key determinants for patients to fulfill the Return-to-Play (RTP) criteria after an anterior cruciate ligament reconstruction (ACLR), in which the muscle size is directly linked to muscle strength. Quadriceps muscle atrophy is unavoidable after ACLR, but the rehabilitation program should increase quadriceps muscle mass. However, despite good rehabilitation compliance, some patient's progress is sub-par and fail to regain muscle mass. Quadriceps muscle atrophy can persist beyond the completion of the rehabilitation program in almost half the patients and the reason behind this is still unknown. This represents an area that requires significant investigation, as quadriceps muscle atrophy and weakness have been shown to be determinants of poor knee function, decreased performance in sports and increased risk of reinjury.

Quadriceps muscle atrophy after ACLR is well documented. This can be due to a decreased ability to regain muscle mass with rehabilitation. Athletes are one of the high-risk groups for vitamin D insufficiencies. Vitamin D deficiency can potentially result in decreased hypertrophy when exercising the muscle, leading to a poorer outcome in rehabilitation. Vitamin D has long been recognized for its effect on musculoskeletal health. It can have a direct effect on muscle hypertrophy by acting on specific vitamin D receptors (VDRs) on myocytes, and sufficient or increased levels of vitamin D in patients have been found to correlate with an increase in the size, number, and strength of muscle fibres. Quadriceps muscle hypertrophy after ACLR is triggered by exercise training, facilitated by diet and a number of intrinsic factors. As the rehabilitation programs and diets are similar in patients with varying extents of quadriceps muscle atrophy, individual responses (intrinsic factors) to exercise training may account for the resulting persistent quadriceps muscle atrophy. In this study, the investigators hypothesize that the deficiency of vitamin D may contribute to persistent quadriceps atrophy and weakness.

With a stringent double-blinded randomized-controlled-trial (RCT) research design, our proposal will then address the research questions: 'Does vitamin D supplements improve the vitamin D deficiency status in patients after ACL reconstruction?', and 'Does vitamin D supplements improve quadriceps muscle strength for patients after ACLR?'

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-40 with unilateral ACL injury
2. Sporting injury with a Tegner score of 7
3. Pre-op serum vitamin D level <20 ng/ml
4. 4 months post-ACLR with serum Vitamin D level remained <20ng/ml
5. LSI for quadriceps strength <70% of contralateral leg at 4-month isokinetic assessment
6. Both knees without history of injury/prior surgery

Exclusion Criteria:

1. Concomitant bone fracture, major meniscus injury or full-thickness chondral injuries requiring altered rehabilitation program post-operatively
2. Pre-operative radiographic signs of arthritis
3. Metal implants that would cause interference on MRI
4. Non-HS graft for ACLR
5. Patient non-compliant to the rehabilitation program
6. Regular sunbed users

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2028-03-17 (Estimated); Study Completion 2029-09-17 (Estimated)

PRIMARY OUTCOMES:
Change of Isokinetic muscle strength | Pre operation, 4-, 6- 8- and 12months post operation
  The dynamometer (Biodex System 4, Biodex Medical Systems Inc., New York, USA) will be used for measuring Isokinetic muscle strength in N. Subjects will perform a standardized warm-up exercise (5 min cycling) followed by the test. Concentric/concentric contractions of knee extension/flexion will be tested at 60°/s and 180°/s. Subjects will be seated on the dynamometer chair with their hips flexed to 85°.
Change of Biochemical Assays | Pre operation, 4-, 6- 8- and 12months post operation
  Blood samples will be taken under non-fasting conditions. Serum / plasma obtained will be immediately stored at -80°C until analysis. Serum 25(OH) Vit-D assay: Serum 25(OH)Vit-D levels will be measured by commercial 25(OH) Vitamin D ELISA kit (Abcam ab213966) according to the manufacturer's instruction, providing the quantitative determination of 25(OH) Vitamin D3 and 25(OH) Vitamin D2. Sensitivity: 1.98 ng/ml (Range: 0.5 ng/ml - 1010 ng/ml).

SECONDARY OUTCOMES:
MRI Muscle thickness | 4- & 8- months post operation
  Muscle volumes of quadricep muscle are measured using a 1.5 or 3.0 Tesla MRI Scanner. Axial (3mm thick cut) T1W images are obtained from the anterior superior iliac supine (ASIS) to patella. Quadriceps muscles were manually outlined in each axial slice. Muscle volume was calculated by summing all of the slice-multiplied by slice thickness. The quality of the muscle is assessed by analyzing the fat content of the muscle mass using technique that has been reported by Reeder et al (6). Bilateral legs will be performed before the start of the vitamin supplementation (4 months post-op) and with the injured side repeated after the completion of the 16-weeks supplementation (8 months postop).The uninjured side will be used as reference for 'normal volume'.
Ultrasound imaging muscle thickness | Pre operation, 4-, 6- 8- and 12months post operation
  The Aixplorer® ultrasound system and a linear transducer probe with a bandwidth of 2-10 MHz were used to measure the muscle thickness of Vastus Medialis (VM), Vastus Lateralis (VL), and Rectus Femoris (RF) on both the injured and uninjured leg. Participants laid supine on a treatment table for the assessment. A measuring tape was used to locate VM, VL, RF and the patella by palpation, consequently marked with a pen for reference. RF was marked at 1/2 of the distance from the anterior superior iliac spine (ASIS) to the superior pole of the patella, VM was located at 1/5 of the distance away from the midpoint of the medial patella border to the ASIS, and VL was noted at 1/3 of the distance from the midpoint of the lateral patella border to the ASIS. After locating the anatomical points, excess contact gel was applied on these points. The transducer probe was aligned in the transverse plane and moved along the entire muscle bundle to capture a view of the VM, VL and RF.
Passive Knee laxity | Pre operation, 4-, 6- 8- and 12months post operation
  To measure anterior-posterior knee laxity, the KT-1000 knee ligament arthrometer (MEDmetric Corp, San Diego, CA, USA) will be used. A manual force test will be applied until a 30lb sound signal is activated. Three trials will be performed. A side difference of 3 mm above is considered clinically relevant.
Change of BMI Anthropometric Measurement | Pre operation, 4-, 6- 8- and 12months post operation
  Body Mass Index (BMI) in kg/m^2 would be calculated by the measured height and weight at 4 months post ACLR before vitamin D supplements, during the eighth week of vitamin D supplements, after the completion of 16 weeks vitamin D supplements, and 12-months post-operation.
Ground reaction force | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  The Kinetic variables including vertical and horizontal ground reaction force (GRF) will be evaluated by a synchronized force plate at the centre of the capture volume at 1000Hz.
Knee Joint moments | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  The kinematics will be assessed by the skin marker-based motion analysis system with the lower-body marker setup followed the OSTRC standard using 16-camera and 16 reflective skin marker during the single leg squat and single leg hop test.
Single leg hop distance | 4weeks, 8 weeks and 8 months after the commencement of intervention
  The average of single leg hop distance in cm with three attempts will be measured during the single leg hop test.
Visual Analogue Scale | Before and immediate after 1st - 16th of PEMF treatment
  The subjective measurement for chronic and acute pain will be recorded by the Visual Analogue Scale (VAS). VAS consists of a 10-cm line which represents the continuum between "painless" and "worst pain from 0 cm to 10 cm. The subject will be asked to draw a mark of it before and after each PEMF treatment session.
Tegner activity score | Pre operation, 4-, 6- 8- and 12months post operation
  This is an activity level scaled from 1 (low activity) to 10 (high activity).
International Knee Documentation Committee | Pre operation, 4-, 6- 8- and 12months post operation
  Consists of 10 questions on symptoms and activity ranging from 0 to 100 where 100 implies perfect knee function.
Lysholm knee scoring system | Pre operation, 4-, 6- 8- and 12months post operation
  Consists of eight items, total score ranging from 0 to 100 where higher scores indicate a better outcome with fewer symptoms or disability.
International Physical Activity Questionnaire | Pre operation, 4-, 6- 8- and 12months post operation
  The level of physical activities during the past 7 days will be evaluated with a validated Chinese version of the quantitative physical activity questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers

REFERENCES:
- [Derived] Ong MT, Lu X, Choi BC, Wan SW, Wang Q, Man GC, Lui PP, Fong DT, Mok DK, Yung PS. Vitamin D as an intervention for improving quadriceps muscle strength in patients after anterior cruciate ligament reconstruction: study protocol for a randomized double-blinded, placebo-controlled clinical trial. Trials. 2024 Apr 11;25(1):251. doi: 10.1186/s13063-024-08094-w. PMID 38605374

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT05174611/Prot_000.pdf
  • Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT05174611/ICF_001.pdf